CLINICAL TRIAL: NCT00463827
Title: Effect of Statins on Asthma Control and Airway Inflammation in Smokers With Asthma: a Randomised Controlled Double-blind Parallel Group Study
Brief Title: Effect of Statins on Asthma Control in Smokers With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NHS Greater Clyde and Glasgow (Other)
Collaborators: University of Glasgow (Other); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Neil Thomson, Professor of Respiratory Medicine, NHS Greater Clyde and Glasgow
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR 003
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Asthma; COPD; Smoking
Keywords: asthma; smokers; statin; atorvastatin; randomised; placebo; cigarette; blind; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Smoking | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Atorvastatin 40
  Interventions: Drug: Atorvastatin
- placebo (Placebo Comparator): matched placebo
  Interventions: Drug: matched placebo

INTERVENTIONS:
Drug: Atorvastatin
  Arms: 2
Drug: atorvastatin — atorvastatin 40mg
  Arms: 2
Drug: matched placebo — Matched placebo
  Arms: placebo

SUMMARY:
Asthma is a chronic inflammatory condition of the lungs.

There is evidence that cigarette smoking can make asthma symptoms worse and that smokers with asthma do not respond as well to standard therapies as non-smokers.

Statins are drugs which are already used to lower cholesterol. They have also been shown to have some anti-inflammatory properties.

In this trial the investigators will give a randomised group of smokers Atorvastatin and the remaining group a placebo or blank tablet. The investigators will then monitor patients' responses in terms of peak flow data, symptom diaries, questionnaires and breathing tests.

DETAILED DESCRIPTION:
Despite several studies, which have shown that smokers with asthma have more severe symptoms, accelerated decline in lung function and diminished response to treatment with inhaled and oral corticosteroids, more than 25% of asthmatics continue to smoke. Smoking cessation advice is often ineffective.

Statins are used as cholesterol lowering agents, however, there is now also evidence that they have additional anti-inflammatory effects which may be useful in treatment of smokers with asthma.

This is a randomised placebo controlled double-blind parallel group study.

Following screening to assess suitability for the study, patients will be randomised to treatment with either Atorvastatin 40mg or placebo (blank tablet)for 8 weeks.

After 4 weeks of treatment, all patients will be commenced on a low dose inhaled corticosteroid for the remainder of the study to assess whether treatment with statins can overcome steroid resistance in smokers with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma for more than 1 year
* Symptomatic asthma
* Smoker with greater than 5 pack year history
* On short acting bronchodilator only- although may have medication weaned if stable

Exclusion Criteria:

* Ex-smokers or non-smokers
* Patients already on statin therapy
* Unstable asthma
* Previous statin sensitivity or myopathy or myositis
* On any medications known to interact with statins

Note separate entry criteria for pilot study of COPD patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in peak flow data | 4 weeks

SECONDARY OUTCOMES:
sputum cell counts | 4 weeks and 8 weeks
spirometry | 4 weeks and 8 weeks
airway responsiveness to methacholine | 4 weeks and 8 weeks
symptom scores | 4 weeks and 8 weeks
Exhaled and alveolar NO | 4 weeks and 8 weeks
Exacerbation rates | 4 and 8 weeks
immunological tests in blood | 4 and 8 weeks
ACQ score | 4 and 8 weeks
AQLQ score | 4 and 8 weeks
Safety issues | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil Thomson, FRCP, Principal Investigator — University of Glasgow
Locations (1):
- Gartnavel General Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Braganza G, Chaudhuri R, McSharry C, Weir CJ, Donnelly I, Jolly L, Lafferty J, Lloyd SM, Spears M, Mair F, Thomson NC. Effects of short-term treatment with atorvastatin in smokers with asthma--a randomized controlled trial. BMC Pulm Med. 2011 Apr 7;11:16. doi: 10.1186/1471-2466-11-16. PMID 21473764
- See also: Unit website — http://www.gla.ac.uk/departments/immunology/index.html